CLINICAL TRIAL: NCT04295707
Title: Accrued Effect of Orthokeratology for Myopia Control in Children and the Effectiveness of Myopia Control Using an Innovative Orthokeratology Modality. Experiment 1. Effect in Existing Ortho-k Wearers
Brief Title: Monthly Replacement Orthokeratology for Myopia Control in Existing Lens Wearers
Acronym: MR1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Menicon Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Pauline Cho, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20190926004-1
Record Dates: First submitted 2020-02-29; First posted 2020-03-04 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Myopic Progression
Keywords: Myopia progression; Orthokeratology; Replacement modality; Surface deposits

STUDY DESIGN:
Intervention Model Description: All subjects will be randomly assigned to use monthly or yearly replacement orthokeratology for a period of 24 months. Subjects on monthly replacement modality will be randomly assigned to normal cleaning and intensive cleaning groups. Subjects in normal cleaning group will be provided with complimentary contact lenses solutions for daily cleaning and disinfection. In addition to the daily procedures for lens case, subjects in the intensive cleaning group will be required to perform weekly protein removal.
  Intensive cleaning is indicated for yearly replacement modality, thus, no randomization of care procedures in this group.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor was responsible for measuring the axial length and was unaware of the replacement modality of intervention used by the subjects. Another independent examiner will be responsible for grading surface coating from the images taken without disclosure of the information on the cleaning procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Monthly replacement orthokeratology without protein removal (Experimental): Subjects will be required to perform daily cleaning for the monthly replacement orthokeratology lenses
  Interventions: Device: orthokeratology
- Monthly replacement lenses with weekly protein removal (Active Comparator): Subjects will be required to perform both daily cleaning and weekly protein removal for the monthly replacement orthokeratology lenses
  Interventions: Device: orthokeratology; Device: Menicon Progent A+B
- Yearly replacement lenses with weekly protein removal (Active Comparator): Subjects will be prescribed with orthokeratology lenses which will be replaced at least every 12 months during the study period. They will be required to perform both daily cleaning and weekly protein removal for their lenses.
  Interventions: Device: orthokeratology; Device: Menicon Progent A+B

INTERVENTIONS:
Device: orthokeratology — Nightly wear of orthokeratology lenses to correct vision in the daytime
  Other Names: ortho-k; Menicon Z Night lenses; Menicon Z Night Toric lenses; corneal reshaping therapy
Device: Menicon Progent A+B — Menicon Progent A+B is a commercially available protein remover for rigid lenses. It has received FDA clearance and been launched in Hong Kong for over a decade. The product contains two separate sterile solutions, one with sodium hypochlorite and the other with potassium bromide. By mixing the two solutions in a special vial, it can clean and remove protein deposits on the lenses. Parents of subjects assigned to use weekly protein remover will be required to soak the cleansed lenses in the solution mixture for not more than 30 mins every week. All lenses must be rinsed thoroughly with saline and cleansed with daily cleaner again before daily disinfection.
  Other Names: Menicon Progent Protein Remover for Rigid Gas Permeable Contact Lenses
  Arms: Monthly replacement lenses with weekly protein removal; Yearly replacement lenses with weekly protein removal

SUMMARY:
The two-year prospective study aims at investigating the benefits of frequent replacement (monthly) orthokeratology lenses in myopia control in terms of effectiveness in control and prevention of ocular complications. The secondary objective will be investigating the use of weekly protein removal system in monthly replacement modality orthokeratology lenses on surface deposit.

DETAILED DESCRIPTION:
This is a two-year randomized trial. Existing orthokeratology lens wearers (aged 8-13 years), who have completed a 2-year myopia control using orthokeratology, will be recruited and monitored for another two years. Eligible subjects will be randomly assigned to monthly or yearly replacement modality. Axial elongation and ocular conditions will be compared between the monthly and yearly replacement groups.

Subjects on monthly replacement lenses will be randomly assigned to normal cleaning and intensive cleaning groups. Subjects in normal cleaning group will be provided with complimentary contact lenses solutions for daily cleaning and disinfection. In addition to the daily procedures for lens case, subjects in the intensive cleaning group will be required to perform weekly protein removal. All subjects on yearly replacement lenses will be required to performed intensive cleaning such that they will follow normal daily cleaning and disinfection as well as weekly protein removal.

ELIGIBILITY:
Inclusion Criteria:

* Aged 8-15 years
* Have completed a two-year myopia control study using ortho-k
* Normal ocular and general condition and not on medication which may contraindicate ortho-k lens wear
* Pre-ortho-k refractive sphere between -0.75 to -4.00 DS, refractive cylinder ≤ -1.50 DC and anisometropia ≤ -1.00 D
* Best correctable vision better than 0.08 logMAR in the worse eye
* Normal binocular function and accommodative status

Exclusion Criteria:

* Strabismus at distance or near
* Contraindication for ortho-k lens wear
* Prior history of ocular surgery, trauma, or chronic ocular disease
* Systemic or ocular conditions that may interfere refractive development
* Systemic or ocular conditions that may interfere tear quality and contact lens wear
* Poor response to the use of study lenses
* Poor compliance to test procedures
* Poor compliance to the use of ortho-k lenses (e.g. use of solution, use of lenses)
* Poor compliance to follow-up schedule

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2020-03-11 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Axial elongation in 2 years | 2 years
  Cycloplegic examination of the eyeball length using IOLMaster every 6 monthly
Back Surface Lens Deposits | Every month up to 12 months
  Surface deposits will be graded using a 4-point scale: 0=no deposit; 1=mild; 2=moderate; 3=severe

SECONDARY OUTCOMES:
Number of participants with serious adverse effects in 2 years | 2 years
  Number of subjects with serious adverse effects of the cornea, the palpebral, bulbar and tarsal conjunctiva in 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Cho, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Optometry, The Hong Kong Polytechnic University, Kowloon, Hong Kong

REFERENCES:
- [Background] Lee YC, Wang JH, Chiu CJ. Effect of Orthokeratology on myopia progression: twelve-year results of a retrospective cohort study. BMC Ophthalmol. 2017 Dec 8;17(1):243. doi: 10.1186/s12886-017-0639-4. PMID 29216865
- [Background] Stapleton F, Carnt N. Contact lens-related microbial keratitis: how have epidemiology and genetics helped us with pathogenesis and prophylaxis. Eye (Lond). 2012 Feb;26(2):185-93. doi: 10.1038/eye.2011.288. Epub 2011 Dec 2. PMID 22134592
- [Background] Cho P, Cheung SW. Retardation of myopia in Orthokeratology (ROMIO) study: a 2-year randomized clinical trial. Invest Ophthalmol Vis Sci. 2012 Oct 11;53(11):7077-85. doi: 10.1167/iovs.12-10565. PMID 22969068
- [Background] Hiraoka T, Kakita T, Okamoto F, Takahashi H, Oshika T. Long-term effect of overnight orthokeratology on axial length elongation in childhood myopia: a 5-year follow-up study. Invest Ophthalmol Vis Sci. 2012 Jun 22;53(7):3913-9. doi: 10.1167/iovs.11-8453. PMID 22577080
- [Background] Cheung SW, Boost MV, Cho P. Pre-treatment observation of axial elongation for evidence-based selection of children in Hong Kong for myopia control. Cont Lens Anterior Eye. 2019 Aug;42(4):392-398. doi: 10.1016/j.clae.2018.10.006. Epub 2018 Oct 24. PMID 30366778